CLINICAL TRIAL: NCT04757415
Title: Effects of Gluteal Activation With or Without Traction Straight Leg Raise Technique Among Patients of Sacroiliac Joint Syndrome
Brief Title: Gluteal Activation With or Without Traction Straight Leg Raise Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/LHR/20/0103 Farzana Saqib
Record Dates: First submitted 2021-02-05; First posted 2021-02-17 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: SIJ - Sprain of Sacroiliac Joint; Weakness, Muscle; Tightness of Back Muscles
Keywords: Gluteal activation; Straight leg raise hamstring technique; Sacroiliac joint pain
MeSH Terms: conditions — Muscle Weakness

STUDY DESIGN:
Who Masked: Participant
Masking Description: single
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traction straight leg raise technique for hamstring. (Experimental): Experimental group underwent conventional physiotherapy treatment (hot pack) followed by five main gluteal activation exercises three in first five sessions and rest two in remaining five sessions along with traction straight leg raise technique. Each session took 30 minutes . Participants were treated 10 times over a 5 week period with 2 treatment sessions per week. Pre and Post treatment readings were taken in 1st and 10th session over a 5 week period respectively. Assessment was done via Numeric pain rating scale and sphygmomanometer for assessing pain intensity and muscle strength of gluteus maximus.
  Interventions: Other: Traction straight leg raise technique for hamstring
- Gluteal activation exercises (Experimental): Experimental group underwent conventional physiotherapy treatment (hot pack) followed by five main gluteal activation exercises three in first five sessions and rest two in remaining five sessions. Each session took 30 minutes . Participants were treated 10 times over a 5 week period with 2 treatment sessions per week. Pre and Post treatment readings were taken in 1st and 10th session over a 5 week period respectively. Assessment was done via Numeric pain rating scale and sphygmomanometer for assessing pain intensity and muscle strength of gluteus maximus.
  Interventions: Other: Gluteal activation exercises,Hotpack

INTERVENTIONS:
Other: Traction straight leg raise technique for hamstring — traction straight leg raise technique is used along with gluteal exercises
  Arms: Traction straight leg raise technique for hamstring.
Other: Gluteal activation exercises,Hotpack — only gluteal activation exercises were performed without traction straight leg raise technique
  Arms: Gluteal activation exercises

SUMMARY:
This study was a Randomized clinical trial conducted to determine the Effects of gluteal activation with or without traction straight leg raise technique among patients of sacroiliac joint syndrome so that in future this study will be helpful for other clinician to determine that how much gluteal activation is important in low back pain or sacroiliac joint syndrome, and how it affects our sling system.

DETAILED DESCRIPTION:
Non Probability Convenient sampling was done . Patients following eligibility criteria from Sports and Spine Professionals ,Lahore were considered. Sample size was calculated with Epi tool calculator. 38 Participants were randomly allocated in two groups equally via convenient sampling method. Baseline assessment was done initially. Group A was given gluteal activation exercises with traction straight leg raise technique for hamstring and Group B was gluteal activation exercises without traction straight leg raise technique for hamstring. Duration of research was almost 6 months. Patient will undergo 10 treatments in five weeks. Each session will take 30 minutes. Pre and Post treatment readings were taken in 1st and 10th session over a 5 week period respectively. Assessment was done via sphygmomanometer and numeric pain rating scale for assessing muscle strength of gluteus maximum and pain levels respectively. All participants were provided written informed consent prior to commencement of the procedures. They were free to quit the treatment at any stage of research. Data was analyzed by using SPSS version 23.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with LBP below the level of L5,
2. With pain over the posterior aspect of SI joint around posterior superior iliac spine and buttock with or without above knee leg pain.
3. Females only

Exclusion Criteria:

1. Had radicular pain with neurological (sensory or motor) deficits,
2. Had a history of spinal surgery, spinal, pelvic, or lower extremity fracture; hospitalization for trauma or motor vehicle accident;
3. Hip or knee dysfunctions;
4. Pregnancy;
5. Any systemic disease such as arthritis, tuberculosis, liver, or kidney failure
6. Subjects with leg length discrepancies, because of its potential effect on hamstring muscle length were also excluded. -

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — females above 40years having sacroiliac joint syndrome
Enrollment: 38 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Change of muscle strength of gluteus maximum by "Sphygmomanometer" | Baseline at 1st session on 1st week,at 10th sessions on 5th week
  change in strength of gluteal muscle was checked at 1st session and then follow up at end of 10th session

SECONDARY OUTCOMES:
change in pain by "Numeric Pain rating Scale" | Baseline at 1st session on 1st week , at 10th session on 5th week
  change in pain intensity was checked at 1st session and then follow up at end of 10th session

CONTACTS AND LOCATIONS:
Overall Officials: Rabiya Noor, PhD, Principal Investigator — Riphah International University
Locations (1):
- Riphah IU, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Massoud Arab A, Reza Nourbakhsh M, Mohammadifar A. The relationship between hamstring length and gluteal muscle strength in individuals with sacroiliac joint dysfunction. J Man Manip Ther. 2011 Feb;19(1):5-10. doi: 10.1179/106698110X12804993426848. PMID 22294848
- [Background] Added MAN, de Freitas DG, Kasawara KT, Martin RL, Fukuda TY. STRENGTHENING THE GLUTEUS MAXIMUS IN SUBJECTS WITH SACROILIAC DYSFUNCTION. Int J Sports Phys Ther. 2018 Feb;13(1):114-120. PMID 29484248
- [Background] Feeney DF, Capobianco RA, Montgomery JR, Morreale J, Grabowski AM, Enoka RM. Individuals with sacroiliac joint dysfunction display asymmetrical gait and a depressed synergy between muscles providing sacroiliac joint force closure when walking. J Electromyogr Kinesiol. 2018 Dec;43:95-103. doi: 10.1016/j.jelekin.2018.09.009. Epub 2018 Sep 22. PMID 30267967
- [Background] Chance-Larsen K, Littlewood C, Garth A. Prone hip extension with lower abdominal hollowing improves the relative timing of gluteus maximus activation in relation to biceps femoris. Man Ther. 2010 Feb;15(1):61-5. doi: 10.1016/j.math.2009.07.001. Epub 2009 Aug 12. PMID 19679506